CLINICAL TRIAL: NCT04401306
Title: Remote Training in Laparoscopy: A Randomized Trial Comparing Home-based Self-regulated Training to Centralized Instructor-regulated Training.
Brief Title: Remote Training in Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other); North Denmark Region (Other Government); KARL STORZ Endoscopy Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: sbs_au235143
Record Dates: First submitted 2020-05-13; First posted 2020-05-26 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2020-05

CONDITIONS: Educational Problems; Surgery
Keywords: Education; Simulation; Surgery; Transfer; Self-regulated learning; Gynecology; Urology; Laparoscopy; Home

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-regulated simulation training (Experimental)
  Interventions: Other: Home-based self-regulated simulation training (SRST)
- Instructor-regulated simulation training (Active Comparator)
  Interventions: Other: Centralized instructor-regulated simulation training (IRST)

INTERVENTIONS:
Other: Home-based self-regulated simulation training (SRST) — Participants allocated to the SRST arm train basic laparoscopic skills at home. Participants train by themselves using a portable box training model (BT). Training is conducted and structured through an online application-based training platform. Training is instructed by online instructional videos and texts. The BT is connected to a laptop and the participants can submit videos of their training exercises for assessment through the online training platform.
  Arms: Self-regulated simulation training
Other: Centralized instructor-regulated simulation training (IRST) — Participants allocated to the IRST arm train basic laparoscopic skills at the simulation centre. Participants train on a portable box training model (BT). Training is structured through an online application-based training platform and facilitated and instructed by surgical specialists. The BT is connected to a laptop and the participants can submit videos of their training exercises for assessment through the online training platform.
  Arms: Instructor-regulated simulation training

SUMMARY:
The study is a prospective, randomized comparative study using a mixed methods design. The primary objective is to compare the effect of self-regulated simulation training (SRST) to instructor-regulated simulation training (IRST) in basic laparoscopic skills. The study population is first-year trainees in the specialties General Surgery, Urology and Obstetrics and Gynaecology within the postgraduate training region of northern Denmark. 46 first-year trainees will be randomized into two groups, one receiving SRST and one receiving IRST in basic laparoscopic skills.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a medical doctor
* Participant is a first-year trainee in abdominal surgery, urology, or gynaecology and obstetrics.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Performed > 50 lap procedures prior to enrollment
* participated in training programs provided by the former course provider in the postgraduate training region of northern Denmark

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Mean time for laparoscopic skills test (LASTT). | 0-7 months
  Laparoscopic skills testing models (pre-test, post-test and retention-test). Scoring based on mean timing of 3 consecutively performed exercises (0-180 secs). Low time-scores are better than high time scores.

SECONDARY OUTCOMES:
Test-score SUTT | 1-7 months
  Laparoscopic knot tying testing model (post-test and retention test). Blinded outcome assessor. Score based on timing and quality of sutures and stitches (score range -2 to 18). High score is better than low score.
Training time | 6-8 weeks
  Accumulated raw training time (mins)
Training distribution | 6-8 weeks
  Number of training sessions
Pass-rates | 6-8 weeks
  Pass/failure of proficiency-based training program (binary)

OTHER OUTCOMES:
Interview | 0-3 months
  Qualitative data: Semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Sigurd B Sloth, MD, PhD fellow, Principal Investigator — Centre for Health Sciences Education, Aarhus University, Denmark
Locations (1):
- Centre for Health Sciences Education, Aarhus University, Aarhus, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided